CLINICAL TRIAL: NCT04476823
Title: Practice in Clinical and Molecular Thoracic European Pathology Laboratories During the COVID-19 Pandemic.
Brief Title: European Pathology Laboratories and COVID-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20labocovid01
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Clinical Practice During the COVID-19 Crisis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Activity — The questionnaire had requested information on the biosafety organization, impact of the COVID-19 crisis on the clinical and molecular pathology and the biobanking activity in thoracic pathology, on the research activity associated with the COVID-19, and on the educational and training organization. It requested the different needs planned by the different laboratories following the COVID-19 crisis and finally the consequence of this latter on the health and virological status of the staff members.

SUMMARY:
The infectivity of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), notably when handling human samples, remains poorly understood, as well as the impact of the COVID-19 pandemic in routine clinical and molecular pathology practice, and for personal working in pathology laboratories. This study evaluates the consequences of the COVID-19 crisis in clinical and molecular pathology laboratories in Europe mostly those orientated for diagnosis of thoracic diseases.

ELIGIBILITY:
Inclusion Criteria:

* laboratories following the COVID-19 crisis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathology laboratories belonging to the Lung working group of the European Society of Pathology and to additional European pathology laboratories expert in thoracic diseases
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Activity | 1 day
  The activity of the pathology laboratories has been compared for a same period (from the 15th of March 15 to the 31th of May) in 2019 and in 2020

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France